CLINICAL TRIAL: NCT00050232
Title: Safety and Efficacy of AVP-923 for Pseudobulbar Affect in Multiple Sclerosis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avanir Pharmaceuticals (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 02-AVR-106
Record Dates: First submitted 2002-12-02; First posted 2002-12-03 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Multiple Sclerosis
Keywords: Pseudobulbar Affect; Uncontrolled; Laughing; Crying
MeSH Terms: conditions — Multiple Sclerosis; Laughter; Crying | interventions — dextromethorphan - quinidine combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AVP-923

SUMMARY:
Pseudobulbar Affect is a condition characterized by frequent episodes of laughing and crying out of proportion. Other terms used to describe this condition include emotional lability, emotionalism, emotion incontinence, emotional discontrol, excessive emotionalism and pathological laughing and crying. AVP-923 is a new experimental drug that may assist in the reduction of uncontrolled episodes. This study will test the safety and efficacy of AVP-923 in the treatment of MS patients suffering from pseudobulbar affect.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 68 years of age
* Confirmed diagnosis of Multiple Sclerosis
* Clinical history of pseudobulbar affect

Exclusion Criteria:

* Sensitivity to quinidine or opiate drugs
* Recent diagnosed within 2 months with Multiple Sclerosis
* Patient on anti-depressants
* Patient with liver or kidney disease
* Patient with hypotension

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96
Dates: Start 2002-12; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
emotional control

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Barrow Neurological Institute, Phoenix, Arizona
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Neurological Associates, Fort Lauderdale, Florida
  - Neurology & Headache Specialist of Atlanta, L.L.C., Decatur, Georgia
  - Radiant Research Alexian Brothers, Elk Grove Village, Illinois
  - Consultants in Neurology LTD, Northbrook, Illinois
  - Advanced Neurology Specialists, Great Falls, Montana
  - Neurological Associates, P.C., Lincoln, Nebraska
  - Upstate Clinical Research, Albany, New York
  - DENT Neurologic Group L.L.P., Amherst, New York
  - Hospital for Joint Diseases - MS Care Center, New York, New York
  - Institute for Human Performance, Syracuse, New York
  - Raleigh Neurology Associates, P.A., Raleigh, North Carolina
  - NeuroCare Center, Inc., Canton, Ohio
  - Leheigh Valley Neurosciences and Pain Research Center, Allentown, Pennsylvania
  - Westmorland Neurology, Greensburg, Pennsylvania
  - Neurological Associates of Delaware Valley, Upland, Pennsylvania
  - FACH-UHC Department of Neurological Services, Burlington, Vermont
  - Swedish Medical Center, Seattle, Washington
  - Neurology and Neurosurgery Associates of Tacoma, Tacoma, Washington

REFERENCES:
- [Result] Panitch HS, Thisted RA, Smith RA, Wynn DR, Wymer JP, Achiron A, Vollmer TL, Mandler RN, Dietrich DW, Fletcher M, Pope LE, Berg JE, Miller A; Psuedobulbar Affect in Multiple Sclerosis Study Group. Randomized, controlled trial of dextromethorphan/quinidine for pseudobulbar affect in multiple sclerosis. Ann Neurol. 2006 May;59(5):780-7. doi: 10.1002/ana.20828. PMID 16634036
- See also: National Multiple Sclerosis Society — http://www.nmss.org